CLINICAL TRIAL: NCT00638261
Title: Adalimumab in Primary Combination With UVB-311nm Half-side Phototherapy in Patients With Psoriasis
Brief Title: Primary UVB-311nm and Adalimumab in Psoriasis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Peter Wolf, MD, Professor of Bioimmunotherapy, Medical University of Graz
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-134 ex 07/08
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Psoriasis
Keywords: Psoriasis; Biologic; Adalimumab; Narrow-band UVB; phototherapy; half-side comparison
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- left/right (Other): left or right body side
  Interventions: Radiation: UVB-311nm

INTERVENTIONS:
Radiation: UVB-311nm — UVB-311nm radiation given 3 times a week to one randomized body-half
  Other Names: narrow-band UVB radiation

SUMMARY:
Adalimumab, a fully human anti-tumor necrosis factor (TNF) monoclonal antibody has been approved for the treatment of moderate to severe psoriasis. However, in a portion of cases adalimumab does not induce reduction of psoriasis area and severity index (PASI) of 75% or greater, now being considered as gold standard for treatment efficacy. In this study we aim to determine in a randomized half-side comparison whether initial narrowband UVB-311nm phototherapy accelerates and improves the clearance of skin lesions in adalimumab-treated patients.

DETAILED DESCRIPTION:
Patients with moderate to severe psoriasis who are scheduled to receive a standard treatment course of adalimumab (loading dose of 80 mg and thereafter 40 mg s.c. biweekly) are exposed to UVB-311nm phototherapy on a randomized body half (left or right; head exempt) 3 x per week for six weeks and/or until complete response (defined as reduction in PASI to < 3). PASI score, patient visual analogue score (VAS) for therapeutic response, and patient VAS for severity of skin lesions is assessed weekly; and at follow-up visits at month 3, 6, and 12. Paired Wilcoxon testing for differences in PASI and patient VAS scores is done; Fischer exact test is applied to determine differences in complete remission, PASI reduction > 90%, > 75% and/or 50% between body sites.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis patients who are scheduled for treatment with adalimumab.

Exclusion Criteria:

* Pregnancy or lactation
* History of skin cancer
* Presence of or history of malignant skin tumors
* Dysplastic melanocytic nevus syndrome
* Antinuclear antibodies (ds-DNA, Ro/SSA, La/SSB)
* Autoimmune disorders such as Lupus erythematosus or Dermatomyositis
* Photosensitive diseases such as porphyria, chronic actinic dermatitis, Xeroderma pigmentosum, basal cell nevus syndrome, and others
* General poor health status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Modified PASI (psoriasis area and severity index) | 12 months

SECONDARY OUTCOMES:
Patient visual analogue score (VAS) for therapeutic effect | 12 months
Patient VAS for severity of skin lesions | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz, Austria
Locations (1):
- Medical University of Graz, Department of Dermatology, Graz, Austria